CLINICAL TRIAL: NCT02343666
Title: A Clinical Trial of Gene-Modified Stem Cells to Generate HIV-Resistant Cells in Conjunction With Standard Chemotherapy for Treatment of Lymphoma in Patients With HIV Infection
Brief Title: HIV-Resistant Gene Modified Stem Cells and Chemotherapy in Treating Patients With Lymphoma With HIV Infection
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative closure prior to any enrollments
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2673.00; NCI-2014-02395 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2673; 2673.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); R01HL116217 (NIH)
Record Dates: First submitted 2014-12-30; First posted 2015-01-22 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Human Immunodeficiency Virus 1 Positive; Stage I Adult Hodgkin Lymphoma; Stage I Adult Non-Hodgkin Lymphoma; Stage II Adult Hodgkin Lymphoma; Stage II Adult Non-Hodgkin Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Non-Hodgkin Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Non-Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Carmustine; carmustine, poliferprosan 20 drug combination; Filgrastim; Granulocyte Colony-Stimulating Factor; O(6)-benzylguanine; plerixafor; ferric pyrophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (gene modified HPSC) (Experimental): See Detailed Description.
  Interventions: Biological: C46/CCR5/P140K Lentiviral Vector-transduced Autologous HSPCs; Drug: Carmustine; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: O6-Benzylguanine; Drug: Plerixafor

INTERVENTIONS:
Biological: C46/CCR5/P140K Lentiviral Vector-transduced Autologous HSPCs — Given IV
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Biological: Filgrastim — Given SC
  Other Names: Filgrastim XM02; Filgrastim-sndz; G-CSF; Granix; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim; Zarxio
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: O6-Benzylguanine — Given IV
  Other Names: 6-O-BENZYLGUANINE; O(6)-Benzylguanine
Drug: Plerixafor — Given SC
  Other Names: AMD 3100; JM-3100; Mozobil; SDZ SID 791

SUMMARY:
This pilot phase I trial studies the side effects and best dose of human immunodeficiency virus (HIV)-resistant gene modified stem cells in treating HIV-positive patients who are undergoing first-line treatment for Hodgkin or Non-Hodgkin Lymphoma. Stem cells are collected from the patient and HIV-resistance genes are placed into the stem cells. The stem cells are then re-infused into the patient. These genetically modified stem cells may help the body make cells that are resistant to HIV infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and feasibility of infusing C46/CCR5/P140K lentiviral vector-transduced autologous hematopoietic stem progenitor cells (HSPC) (gene modified, HIV-protected HSPC) after standard first line treatment of lymphoma in patients with HIV infection.

II. To determine the dose of carmustine (BCNU) in combination with O6-benzylguanine (O6BG) that results in selection in vivo of gene-modified HIV resistant cells with minimal toxicity.

III. To estimate the effect of HIV infection on the presence of HIV-resistant blood cells as measured by genetic marking for vector sequences before and after highly active antiretroviral therapy (HAART) interruption.

SECONDARY OBJECTIVES:

I. Evaluate the molecular and clonal composition of gene-modified cells after standard first line treatment.

II. Evaluate the molecular and clonal composition of gene-modified cells after O6BG/BCNU.

III. Determine the correlation between the level of MGMT(P140K) marking with toxicity and response to O6BG/BCNU chemotherapy.

IV. Characterize the toxicity associated with in vivo selection.

V. Describe time to disease progression, progression-free survival, treatment-related mortality, time to neutrophil and platelet recovery, and incidence of infections.

TERTIARY OBJECTIVES:

I. Effect of procedure on the latent HIV reservoir.

II. Effect of procedure on HIV-specific immune reconstitution.

OUTLINE:

MOBILIZATION AND HSPC COLLECTION: Between the second and the last course of planned standard chemotherapy, patients undergo mobilization of peripheral blood stem cells with filgrastim subcutaneously (SC) beginning the day after the last dose of chemotherapy in the previous cycle. If CD34 cell count in peripheral blood at least 24 hours after recovery from nadir is >= 40 CD34 cells/mcL, patients will undergo apheresis collection the next day. If CD34 cell count is < 40 CD34 cells/mcL, plerixafor SC will be administered and patients will undergo apheresis collection the next day. Patients undergo apheresis until a total apheresis product of >= 4.0 x 10^6 CD34+ cells/kg are collected.

STEM CELL INFUSION: Patients receive CD34+ gene-modified C46/CCR5/P140K lentiviral vector-transduced autologous HSPC intravenously (IV) within 2 to 8 days, but no later than 28 days, after completion of the last cycle of first line treatment for lymphoma.

IN VIVO SELECTION WITH O6-BENZYLGUANINE AND CARMUSTINE: Between 28-180 days after infusion of gene-modified HSPC and after hematopoietic recovery from first line treatment, patients with >= 1% and < 10% gene marked cells receive O6-benzylguanine IV over 1 hour, immediately followed by carmustine IV, and followed 7-8 hours later by O6-benzylguanine IV over 1 hour. Treatment continues for an additional course provided that gene marked cells does not meet or exceed 10% of peripheral blood cells and in the absence of unacceptable toxicity.

STRUCTURED TREATMENT INTERRUPTION (STI): Patients achieving >= 10% gene marked cells for 2 consecutive months following infusion of gene-modified HSPC and with CD4+ cell counts and total lymphocyte counts at baseline begin STI of HAART for up to 12 weeks. Patients resume HAART if one of the following criteria occurs: 1) CD4 count < 350 cells/mcL or decline in percent CD4+ cells by > 33% from baseline for three consecutive evaluations; 2) increase in HIV RNA > 100,000 copies/mL on two consecutive evaluations; 3) 12 weeks have passed since discontinuation of HAART; or 4) at the discretion of the infectious disease (ID) consultant or principal investigator (PI).

* If patient is not on an efavirenz-containing regimen, HAART is discontinued simultaneously. If patient is on an efavirenz-containing regimen, patients will switch from efavirenz to an integrase inhibitor for at least 2 weeks and then discontinue HAART simultaneously.

After completion of study treatment, patients are followed up for 2 years, every 6 months for 3 years and then annually for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive
* Stable, continuous antiretroviral treatment, defined as a multi-drug regimen (excluding zidovudine, also known as azidothymidine [AZT], Retrovir) prior to enrollment, as demonstrated by HIV plasma viral load < 50 copies/mL
* Previously untreated non-Hodgkin lymphoma or Hodgkin lymphoma; all stages of disease are allowed; also eligible are patients who have started or completed one or more cycles of treatment as part of a planned first line regimen, or those who have received local radiation or surgery or corticosteroids for disease control
* Planned treatment with standard first line therapy for non-Hodgkin lymphoma (NHL) or Hodgkin lymphoma (HL)
* Karnofsky performance score >= 70%
* Subjects must agree to use effective means to prevent conception from enrollment through completion of the study
* Female subjects: if of child bearing potential, must have negative serum or urine pregnancy test within 7 days of enrollment
* Subjects must be on a prophylactic regimen for Pneumocystis jiroveci pneumonia, or agree to begin such treatment, if CD4+ cell counts are observed to be =< 200/ul in peripheral blood
* Able to understand, and the willingness to give, informed consent for the study

Exclusion Criteria:

* Central nervous system (CNS) lymphoma: CNS involvement by lymphoma, including parenchymal brain or spinal cord lymphoma or known presence of leptomeningeal disease prior to registration
* Patients with renal, hepatic, pulmonary, or cardiac disease that exclude delivery of standard chemotherapy
* Active (uncontrolled) infection requiring systemic antibiotic therapy with antibacterial, antifungal, or antiviral agents (excluding HIV)
* Hepatitis B surface antigen positive
* Hepatitis C virus (HCV) antibody positive and detectable HCV quantitative ribonucleic acid (RNA), with clinical evidence of cirrhosis as determined by the principal investigator
* Requiring active treatment for Toxoplasma gondii infection
* Malignancy other than lymphoma, unless (1) in complete remission and more than 5 years from last treatment, or (2) cervical/anal squamous cell carcinoma in situ or (3) superficial basal cell and squamous cell cancers of the skin
* History of HIV-associated encephalopathy; dementia of any kind; seizures in the past 12 months
* Any perceived inability to directly provide informed consent (note: consent may not be obtained by means of a legal guardian)
* Any concurrent or past medical condition that, in the opinion of the investigator, would exclude the subject from participation
* Patients who have received a vaccine for HIV-1 or any prior gene modified cell product, at any time
* A medical history of noncompliance with HAART or medical therapy
* Pregnant women or nursing mothers
* Use of zidovudine as part of the HAART regimen (a drug substitution for zidovudine at the time of study entry is allowed)
* Known hypersensitivity to any of the products used in the trial - G-CSF (Neupogen, filgrastim), plerixafor (Mozobil), or any components of the chemotherapeutic agents or O6BG/BCNU in vivo selection regimens

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of collection: defined as collection of >= 4.0 x 10^6 CD34+ cells/kg for genetic modification | Up to 28 days after completion of last course of first line treatment for lymphoma
Feasibility of infusion of gene modified cells: defined as engraftment of >= 1% gene modified cells | Up to 28 days after infusion of gene-modified cells to 15 years post-transfusion
  Engraftment of >= 1% gene modified cells.
Feasibility of O6-benzylguanine/carmustine in vivo selection: defined as selection of gene modified cells to a level >= 10% of peripheral blood cells | Up to 180 days after infusion of the gene modified hematopoietic stem progenitor cells
Feasibility of structured treatment interruption: defined as the ability to achieve >= 10% gene modified cell engraftment level and maintain CD4 counts and plasma viremia at levels required for structured treatment interruption eligibility | Up to 18 months following infusion of CD34+ gene modified hematopoietic stem progenitor cells
Presence of confirmed replication competent lentivirus | Up to 15 years
  Any development of confirmed replication competent lentivirus in any patient receiving gene modified cells during the study will be recorded.
Presence of insertional mutagenesis | Up to 15 years
  Confirmed insertional mutagenesis in any patient who received gene modified cells during the study
Safety of infusion of gene modified cells: defined as Common Terminology Criteria for Adverse Events version 4 toxicity >= grade 3 related to the infusion of gene modified cells | Up to 30 days after infusion of CD34+ modified hematopoietic stem progenitor cells
Safety of O6-benzylguanine/carmustine in vivo selection, defined as < 25% of patients developing Common Terminology Criteria for Adverse Events version 4 toxicity >= grade 3 associated with O6-benzylguanine/carmustine administration | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Mazyar Shadman, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States